CLINICAL TRIAL: NCT02382029
Title: The Effectiveness of Acupuncture Versus Clonazepam in the Patients With Burning Mouth Syndrome
Brief Title: Acupuncture Versus Clonazepam in Burning Mouth Syndrome
Acronym: ACUCLONBMS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Vanja Vucicevic Boras, Associate professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UZagreb
Record Dates: First submitted 2015-02-13; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Burning Mouth Syndrome
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Clonazepam; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clonazepam (Active Comparator): Twenty two patients took clonazepam two times a day (0.5 mg) in the morning and after two weeks one tablet (0.5 mg) in the morning and another tablet (0.5 mg) in the evening during the next two weeks.
  Interventions: Drug: Clonazepam
- acupuncture (Experimental): Traditional Chinese acupuncture was performed on 20 participants 3 times during one week for four weeks. Intervention was performed on acupuncture points as follows: the points ST 8 (stomach- tou wei), GB 2, TE 21, SI 19 (small intestine- ting gong), SI 18 (small intestine- quan liao), LI 4 (large intestine-Yuan) on both sides of the body as well as GV 20 (Governing vessel-bai hui).
  Each session lasted half an hour. Sterile acupuncture needles made from surgical stainless steel silicone coated with spring handle were used. The dimensions of the chosen needles were 0.25 in diameter and 30 mm length, inserted at the depth of the 0.5-1 cm. The elicited response was of the type "de qi" accompanied by redness and a feeling of numbness around the needles.
  Interventions: Other: acupuncture

INTERVENTIONS:
Drug: Clonazepam — Active medical treatment for burning mouth syndrome
  Other Names: Rivotril
  Arms: clonazepam
Other: acupuncture — Traditional chinese acupuncture
  Arms: acupuncture

SUMMARY:
Objective: Burning mouth syndrome (BMS) is chronic oral condition characterized with burning symptoms which affects perimenopausal and postmenopausal women. It seems that neuropathy might be the underlying cause of the condition. There are still insufficient data regarding successful therapy. The aim of this study was to compare efficacy of acupuncture and clonazepam in 42 BMS patients (38 women, 4 men), age range 66.7±12 years.

Methods: Patients were randomly divided into two groups. Acupuncture was performed in group I during four weeks, 3 times per week on the points ST 8, GB 2, TB 21, SI 19, SI 18, LI 4 on both sides of the body as well as GV 20, each session lasted half an hour.Group II patients took clonazepam two times a day (0.5 mg) in the morning and after two weeks two tablets (0.5 mg) in the morning and in the evening during the next two weeks. Prior to and one month after either therapy, participants fulfilled questionnaires: visual analogue scale, Beck depression inventory, LANSS pain scale, 36-item short form Health Survey (SF-36) and Montreal Cognitive Assessment (MoCA). Statistical analysis was performed by use of Student t test and Pearson's correlation test. P values lower than 0.05 were considered significant.

DETAILED DESCRIPTION:
This study was approved by Ethical Committee of the School of dentistry in Zagreb. Prior to the study every participant signed informed consent according to the Helsinki II. All patient were recruited from the Department of Oral medicine, School of dentistry in Zagreb.

Patients were randomized by simple randomization method- flipping a coin (heads - acupuncture, tails - clonazepam).

Inclusion criteria were symptoms of burning in the oral cavity with clinically healthy appearance of the oral mucosa. Burning symptoms were continuous throughout the day and lasted for more than 6 months. Some of the patients also had hyposalivation and disturbed taste.

Prior to the either therapy as well as after the therapy (one month after the therapy has finished) every participant fulfilled following questionnaires: visual analogue scale (VAS) which referred to the severity of burning symptoms, Beck depression inventory (BDI), The Leeds assessment of neuropathic symptoms and signs (LANSS) Pain Scale, 36-item short form Health Survey (SF-36) total sum score and Montreal Cognitive Assessment (MoCA).

Arm (I) traditional Chinese acupuncture - performed 3 times during one week for four weeks on the points ST 8 (stomach- tou wei), GB 2, TE 21, SI 19 (small intestine- ting gong), SI 18 (small intestine- quan liao), LI 4 (large intestine-Yuan) on both sides of the body as well as GV 20 (Governing vessel-bai hui) and each session lasted half an hour. We used sterile acupuncture needles from surgical stainless steel silicone coated with spring handle, the dimensiones of the chosen needles were 0.25 in diameter and 30 mm lenght, inserted at the depht of the 0.5-1 cun. The elicited response was of the type "de qi" accompanied by redness and a feeling of numbness around the needles.

Arm (II) Clonazepam - patients took clonazepam two times a day (0.5 mg) in the morning and after two weeks one tablet (0.5 mg) in the morning and another tablet (0.5 mg) in the evening during the next two weeks.

Statistical analysis was performed by use of Student t test and Pearson's correlation test. P values lower than 0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of burning mouth syndrome Clinically normal appearance of oral mucosa Must be able to swallow tablets

Exclusion Criteria:

Oral mucosal lesions Anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 6 months
  Pain intensity measured by the visual analogue scale

SECONDARY OUTCOMES:
The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale | 6 months
  Assessment of neuropathic pain measured by validated instrument (LANSS pain scale)
Cognitive function | 6 months
  Assesment of cognitive function measured by validated instrument ( MoCA cognitive test)
Depression | 6 months
  Assesment of depressive symptoms by use of validated instrument (Beck Depression Inventory)
Quality of life | 6 months
  Assesment of quality of life by validated instrument (Short Forma Health Survey: SF-36)